CLINICAL TRIAL: NCT05933122
Title: Study of the Prevalence of Sexual Dysfunction in Women After Rectal Cancer Surgery and Analysis of the Impact of a Sexologist Intervention
Acronym: RectSexQol
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Limoges (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 87RI22_0006
Record Dates: First submitted 2023-06-09; First posted 2023-07-06 (Actual); Last update posted 2024-12-02 (Actual); Status verified 2024-11

CONDITIONS: Rectal Tumor; Women; Sexuality; Life Quality
Keywords: rectal cancer; women; sexuality; quality of life
MeSH Terms: conditions — Rectal Neoplasms; Sexuality

STUDY DESIGN:
Intervention Model Description: * Cohort called "elsewhere" = cohort without specific care by a sexologist
  * Cohort called "here" = cohort with an intervention by a sexologist
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cohort called "elsewhere" (Sham Comparator): cohort without specific care by a sexologist
  Interventions: Other: standart of care
- Cohort called "here" (Experimental): cohort with an intervention by a sexologist
  Interventions: Other: sexologist consult

INTERVENTIONS:
Other: sexologist consult — in the cohort called "here", after the diagnosis of rectal cancer, patients will be seen by a sexologist before any kind of treatment for rectal cancer. Sexual dysfunctions will be assessed by a sexologist. After the surgery of rectal cancer, the sexologist will see them again to assess sexual dysfunctions after such a management of rectal cancer. If there is any discovery of a sexual dysfunction or aggravation of a previous one or alteration of sexual life, the sexologist will help the patients to improve their sexual quality of life.
  Arms: Cohort called "here"
Other: standart of care — in the cohort called "elsewhere" , patients will be treated according to standards of care, without specific care by a sexologist
  Arms: Cohort called "elsewhere"

SUMMARY:
RectSexQoL is a study aiming at determining the prevalence of female sexual dysfunction after rectal cancer surgery. It has the goal as well to analyse the impact of an intervention given by a sexologist to such patients.

DETAILED DESCRIPTION:
The treatment of rectal cancer is multimodal combining surgery, chemotherapy and radiotherapy. Each therapeutic tool may affect the sexual life of treated patients.

The incidence of sexual dysfunction in patients with rectal cancer varies according to literature from 5 to 88%. This may be due to the lack of a common definition relating to sexual dysfunction making it difficult to compare results. On the other hand, it should be noted that all of the work related to sexual dysfunction after treatment for rectal cancer is mainly interested in men. The sexual well-being of women treated for rectal cancer is based on the assessment and management of their sexual functions as well as that of their overall sexual health in a personalized manner. The establishment of a sexology consultation before and after such a surgical procedure could improve the sexual functions as well as the sexual well-being of these women. The main aim of our study is to evaluate the prevalence of sexual dysfunctions at M-1 (before treatment) in the two cohorts "here" and "elsewhere" in the context of surgery for rectal cancer in females. The second aim will be to determine the impact of sexology consultation in the cohort "here" in comparison to the standart cohort without any intervention called "elsewhere".

ELIGIBILITY:
Inclusion Criteria:

* Women
* Diagnosis of stage I-III rectal adenocarcinoma or rectosigmoid junction with anastomosis less than 15 cm from the anal margin
* Surgical management, preceded or not by Radio-chemotherapy, with restoration of continuity
* Age : over 18
* Proficiency in French or English

Exclusion Criteria:

* Current pregnancy
* Significant cognitive/psychiatric disorders
* Guardianship

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 144 (Estimated)
Dates: Start 2024-04-03 (Actual); Primary Completion 2027-05 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
Number and proportion of women with sexual dysfunction defined as a total FSFI | Month -1
  Number and proportion of women with sexual dysfunction defined as a total FSFI ("Female Sexual Function Index") score greater than 26.55 at Month -1 (before any treatment) in the context of surgery for rectal cancer

SECONDARY OUTCOMES:
Number and proportion of women with sexual dysfunction defined as a total FSFI score greater than 26.55 at Month 6 and Month 12 after usual or specific management in the context of surgery for rectal cancer | Month 12
  Number and proportion of women with sexual dysfunction defined as a total FSFI ("Female Sexual Function Index") score greater than 26.55 at Month 6 and Month 12 after usual ("elsewhere" cohort) or specific management (duration of 6 months) ("here" cohort, including consultations by a sexologist supervising the surgical procedure) in the context of surgery for rectal cancer
Change in the score of the "satisfaction" dimension of the FSFI scale between Month -1, Month 6 and Month 12 | Month 12
  Change in the score of the "satisfaction" dimension of the FSFI scale between Month -1, Month 6 and Month 12
Differences (Month 6 - Month -1 and Month 12 - Month 6) in the score of the "satisfaction" dimension of the FSFI scale (Q14-Q16) between the groups with and without treatment by a sexologist (cohort here vs. elsewhere) | Month 12
  Differences (Month 6 - Month -1 and Month 12 - Month 6) in the score of the "satisfaction" dimension of the FSFI scale (Q14-Q16) between the groups with and without treatment by a sexologist (cohort here vs. elsewhere)

CONTACTS AND LOCATIONS:
Locations (6):
- France (6):
  - Brive Hospital, Brive-la-Gaillarde
  - Les cedres Clinical, Brive-la-Gaillarde
  - Gueret Hospital, Guéret
  - Chenieux clinical, Limoges
  - Limoges University Hospital, Limoges
  - Saint Junien Hospital, Saint-Junien

IPD SHARING:
Plan to Share IPD: No